CLINICAL TRIAL: NCT05611541
Title: The Effect of Health Belief Model-Based Progressive Muscle Relaxation Training on Anxiety and Blood Sugar Levels to Women With Gestational Diabetes: A Randomised Controlled Trial
Brief Title: The Effect of Model-Based PMR Training on Anxiety and Blood Sugar Levels to Women With Gestational Diabetes
Acronym: GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nilüfer Tok Yanık, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10428916
Record Dates: First submitted 2022-09-12; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Anxiety in Pregnancy
Keywords: gestational diabetes; Health Belief Model; Progressive Relaxation Exercise; Anxiety; Blood Sugar
MeSH Terms: conditions — Diabetes, Gestational; Anxiety Disorders | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Using a computer program, the researchers randomly placed pregnant women who received dietary advice into either the intervention group or the control group.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Progressive Muscle Relaxation Training Program; The training was carried out in a single session for 2 hours and a break of 10-15 minutes was given.
  Pregnant women were instructed to perform PMR at least 1 hour after dinner 5 days a week.
  Interventions: Behavioral: Diet therapy, Progressive Muscle Relaxation training, Progressive Muscle Relaxation group
- Control group (Active Comparator): The Progressive Muscle Relaxation Training Program and the Progressive Muscle Relaxation were not applied.
  The pregnant women were asked to continue their normal daily activities for 8 weeks.
  Interventions: Behavioral: The group who received diet therapy and practiced their daily activities.

INTERVENTIONS:
Behavioral: Diet therapy, Progressive Muscle Relaxation training, Progressive Muscle Relaxation group — The group that received Progressive Muscle Relaxation training and applied progressive muscle relaxation for 8 weeks.
  Arms: İntervention group
Behavioral: The group who received diet therapy and practiced their daily activities. — The group who received diet therapy and practiced their daily activities.
  Arms: Control group

SUMMARY:
This research is a randomized controlled experimental study to evaluate the effects of PMR application based on HBM in terms of blood sugar and anxiety levels in women with GDM. 34 pregnant women who applied PMR formed the "intervention group" and 34 pregnant women who did not practice PMR formed the "control group". The intervention group received "Progressive Muscle Relaxation Training". It was determined that there was a statistically significant difference between the last follow-up state anxiety score averages, and the intermediate and final follow-up trait anxiety scores between the intervention and control groups. It was determined that PMR provided a decrease in psychological anxiety levels in pregnant women with GDM, and did not have a positive effect on physiologically fasting, 1 hour postprandial and 2 hour postprandial blood glucose levels. PMR training prepared based on HBM is a method that nurses can perform independently to ensure the psychological well-being of pregnant women with GDM.

DETAILED DESCRIPTION:
Aim: This research is a randomized controlled experimental study that includes evaluation of the effects of PMR based on the SIM model in terms of blood sugar and anxiety levels in women with GDM.

Method: The sample group consisted of 68 pregnant women who were diagnosed with GDM for the first time in the Health Sciences University Antalya Training and Research Hospital Gynecology and Obstetrics Polyclinic. 34 pregnant women who applied PMR constituted the "intervention group" and 34 pregnant women who did not practice PMR constituted the "control group". Data collection was done by the researcher. The "Informed Consent Form", "Pregnant Diagnosis Form", "State-Trait Anxiety Inventory-STAI" were applied to women with GDM in the intervention and control groups before the intervention.

Progressive Muscle Relaxation Training was given to the intervention group. Pregnant women in the intervention group applied PMR 1 hour after dinner, 5 days a week, for 8 weeks. The "International Physical Activity Questionnaire-IPAQ" and "Diet Compliance Questionnaire" were applied to both groups every week for eight weeks.The "State-Trait Anxiety Inventory-STAI" was administered to both groups for interim follow-up 4 weeks after the intervention, and the postprandial 1st hour and 2nd hour postprandial blood glucose values were measured.The "State-Trait Anxiety Inventory-STAI" was administered to both groups for the final follow-up, 8 weeks after the intervention, and the postprandial 1st hour and 2nd hour postprandial blood glucose values were measured.The data in the research were analyzed using the IBM SPSS (Statistical Package for Social Sciences) for Windows 25.0 program.

ELIGIBILITY:
Inclusion Criteria:

* At least 24 weeks of pregnancy,
* 19-45 years old (fertility period),
* no history of diabetes before pregnancy,
* First time diagnosed with GDM,
* Body Mass Index (BMI) at a normal level of 18.5-24.9
* Receiving information about diabetes nutrition during pregnancy from the SBUAEAH Diet Polyclinic.
* Those who do not actively participate in birth preparation classes
* Literate,
* Do not have any barriers to prevent communication (hearing, hearing impairment, etc., use of languages other than Turkish),
* Residing in Antalya city center
* Agreeing to blood glucose measurements by the researcher
* Not using complementary therapies based on mind-body techniques such as acupuncture and massage during the research.

Exclusion Criteria:

* Having multiple pregnancies
* Having a diagnosed disease other than GDM (polyhydramnios, multiple pregnancy, pregnancy-induced hypertension, cardiac problems)
* It consisted of women who did not accept to participate in the research.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Level | Before the intervention
  State-Trait Anxiety Inventory is a Likert-type scale consisting of 20 questions that measures state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Anxiety Level | After the 4-week intervention period.
  State-Trait Anxiety Inventory is a Likert-type scale consisting of 20 questions that measures state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Anxiety Level | After the 8-week intervention period.
  State-Trait Anxiety Inventory is a Likert-type scale consisting of 20 questions that measures state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Fasting blood glucose value | Before the intervention
  Peripheral glucose values are recorded at the morning fasting. Mean fasting blood glucose is defined as <95 mg/dL.
Fasting blood glucose value | After the 4-week intervention period.
  Peripheral glucose values are recorded at the morning fasting. Mean fasting blood glucose is defined as <95 mg/dL.
Fasting blood glucose value | After the 8-week intervention period.
  Peripheral glucose values are recorded at the morning fasting. Mean fasting blood glucose is defined as <95 mg/dL.
Postprandial 1 hour blood glucose value | Before the intervention
  Peripheral glucose values are recorded at the morning 1 hour blood glucose. Mean 1 hour blood glucose is defined as <140 mg/dL.
Postprandial 1 hour blood glucose value | After the 4-week intervention period.
  Peripheral glucose values are recorded at the morning 1 hour blood glucose. Mean 1 hour blood glucose is defined as <140 mg/dL.
Postprandial 1 hour blood glucose value | After the 8-week intervention period.
  Peripheral glucose values are recorded at the morning 1 hour blood glucose. Mean 1 hour blood glucose is defined as <140 mg/dL.
Postprandial 2 hour blood glucose value | Before the intervention
  Peripheral glucose values are recorded at the morning 2 hour blood glucose. Mean 2 hour blood glucose is defined as <120 mg/dL.
Postprandial 2 hour blood glucose value | After the 4-week intervention period.
  Peripheral glucose values are recorded at the morning 2 hour blood glucose. Mean 2 hour blood glucose is defined as <120 mg/dL.
Postprandial 2 hour blood glucose value | After the 8-week intervention period.
  Peripheral glucose values are recorded at the morning 2 hour blood glucose. Mean 2 hour blood glucose is defined as <120 mg/dL.

SECONDARY OUTCOMES:
Weekly physical activity level | 8 weeks
  International Physical Activity Questionnaire (IPAQ) Short Form. The IPAQ consists of a total of seven questions questioning short form walking, moderate-intensity physical activity, vigorous physical activity, and time spent sitting. Total score calculation, metabolic equation (MET) values given to activities (vigorous activity=8 METs, moderate-intensity activity=4 METs, walking=3.3 METs, sitting-=1.5 METs), duration (minutes) and frequency of activities (number of days) multiplied and weekly MET-min scores are obtained. Physical activity levels according to total physical activity score; Those with 0-600 MET-minutes/week are classified as physically inactive, those with 600-3000 MET-minutes/week with low physical activity level, those with over 3000 MET-minutes/week as having adequate physical activity level.
Level of compliance with the weekly diet | 8 weeks
  Diet Compliance Questionnaire is a questionnaire consisting of 7 questions structured by the researcher using the literature to determine the diet compliance status of pregnant women, the reasons for not complying with the diet, the status of skipping meals in the diet and the reasons for skipping meals.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Tok Yanık, Principal Investigator — Ege Üniversitesi Hemşirelik Fakültesi
Locations (1):
- Akdeniz Üniversitesi Hemşirelik Fakültesi, Konyaalti, Antalya, Turkey (Türkiye)